CLINICAL TRIAL: NCT03440268
Title: Prevention of Acute Kidney Injury by N-Acetylcystein in Patients Undergone Cardiac Valve Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Jose Jayme Galvão de Lima, Principal investigator, MD (Nefrologist),PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NAC Valve
Record Dates: First submitted 2018-01-05; First posted 2018-02-22 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Surgery--Complications; Cardiac Valve Disease; Acute Kidney Injury; Oxygen Radical Damage; Post-Op Complication
Keywords: cardiac surgery; post operatory complications; Acute kidney injury; N-acetylcystein
MeSH Terms: conditions — Heart Valve Diseases; Acute Kidney Injury; Postoperative Complications | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: There will be one group placebo/control and one group intervention. The group intervention will receive the medication N AcetylCysteyn (NAC), while the control will receive a placebo
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant of the study won't know what is he receiving (placebo or NAC) and the assessor will not have any contact with the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N Acetyl Cysteine (Experimental): NAC in pre operatory 150mg/kg infusion in 2 hours. NAC during the surgery 50mg/kg in 6 hours. The influence of NAC will be assess in post operatory moment with routine exams
  Interventions: Drug: N Acetyl Cysteine
- Placebos (Placebo Comparator): Saline solution in pre operatory. Saline Solution duing the surgery. The post operatory datas of both groups will be compare
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: N Acetyl Cysteine — Administrate NAC in the pre operatory and intra operatory moments and assess the influence in the outcomes
  Other Names: NAC; experimental
  Arms: N Acetyl Cysteine
Drug: Placebos — These participants will receive a saline solution in pre operatory with the same volume as the experimental group, and this solution will be administrated in 2 hours. During the surgery they will receive a new solution with the same volume of the experimental group, and this solution will be administrated in 6 hours too. The solutions will be covered by an opaque bag, so the participant will not see what is being administrated
  Other Names: control
  Arms: Placebos

SUMMARY:
This is a randomized clinical trial, double-blind, placebo-controlled study with the goal to assess the influence of using N-AcetylCysteyn (NAC) for prevention of AKI (Acute Kidney Injury) in post operatory of valve replacement until their discharge or death

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a serious complication after cardiovascular surgery. Pharmacologic interventions to prevent postoperative AKI have been, in general, unsuccessful. N-Acetylcystein (NAC) is a scavenger of reactive oxygen species that prevents renal dysfunction caused by radiocontrast agents but its ability to prevent AKI in cardiovascular surgery remains controversial. Lack of dose standardization and route of administration contributes to conflicting results in the literature. ln a earlier prospective, double-blind, placebo-controlled study 1 the investigators showed that high-dose NAC reduced the incidence of AKI in patients undergoing coronary artery bypass graft surgery. In this research the investigators aim to validate the results of the abovementioned work in a larger group of patients undergoing cardiac valve replacement, using the same protocol. Methods: This will be a unicentric, prospective, double-blind, placebo-controlled investigation. The Institutional Review Board has already approved the study protocol and all participants will sign a written informed consent. Adult patients of both sex scheduled to undergo elective cardiac valve replacement (aortic and/or mitral) at the Heart Institute, University of São Paulo Medical School, will be considered for inclusion. Exclusion criteria: patients younger than 18 years, dialysis, and participation in other studies, allergy to NAC, active infection, emergency cardiac surgery and malignancies. One-hundred fifty-four patients will be randomly allocated (1:1 ratio) to receive either NAC (Fluimucil, Zambon Laboratories, São Paulo, Brazil) 150 mg/kg in 500 mL 0.9% IV saline in 2 hours, started 2 hours before surgery, followed by NAC 50 mg/kg in 500 mL 0.9% IV saline over 6 hours (NAC group) or 0.9% IV saline (control group) at the same volume. This dose was selected because it is the highest dose sanctioned for clinical use 2 and because it has been shown to reduce the oxidative burst response to Cardiopulmonary Bypass (CPB). Allocation will be based on random computer generated numbers. Patients and investigators will be blinded to treatment assignment. Blood samples will be collected 24 hours before surgery and up to 1 week postoperatively. Serum neutrophil gelatinase associated lipocalin (NGAL) and thiobarbituric acid reactive substances will be determined at the same intervals.2 The primary outcome is the incidence of AKI, as defined by the KDIGO and Acute Kidney Injury Network classification 3 , stages 1, 2, or 3, in the first 72 hours after surgery. The secondary outcomes are death by any cause, cardiovascular events (myocardial infarction, stroke, heart failure, and life-threatening arrhythmia), time in the intensive care unit, time of hospitalization and need of dialysis. The investigators will determine thiobarbituric acid reactive substances to verify if changes in renal function would coincide with changes in oxidative stress and NGAL as an additional marker of renal damage. Patients will be followed up until death or hospital discharge. The renoprotective effect of NAC is attributed to its ability to attenuate the oxidative stress burst associated with cardiac surgery and Cardiopulmonary BYPASS (CPB). The present investigation pretend not only to address this problem, but also to offer evidence that NAC abolishes the increase in circulating reactive oxygen species thus giving a plausible explanation for the renoprotective effect of NAC. Given the clinical relevance of AKI associated to cardiac surgery, lack of dependable methods to prevent that complication and the reduced number of prospective, randomized studies addressing the problem, this work has potential practical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Both sex
* Elective replacement valve (mitral or aortic) procedure

Exclusion Criteria:

* Chronic dialysis patients
* Emergency procedures
* Percutaneous procedures
* Pregnants
* Oncologic patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
NAC and acute kidney injury (AKI) | The participants will be assess in the day before the surgery (baseline), and daily until 7 days of post operatory
  Assess the influence of using NAC in the incidence of AKI by using the Kidney diagnosis improving outcomes (KDIGO) score and Acute kidney injury network (AKIN) score that use the creatinine seric and urine output values to define if we can or not diagnosis acute kidney injury in this pacient. The incidence of AKI will be defined by KDIGO criterea: AKI if creatinine raises up to 1,5 times the baseline, until 7 days. Or if seric creatinine raises 0,3mg/dL up to baseline in 48 hours. Urine output: less than 0,5ml/kg/h for 6-12 hours AKIN criterea: AKI if creatinine raises up to 1,5 times the baseline, until 7 days. Or if seric creatinine raises 0,3mg/dL up to baseline in 48 hours. Urine output: less than 0,5ml/kg/h for 6-12 hours

SECONDARY OUTCOMES:
NAC and kidney replacement therapy (KRT) | From the post operatory until the necessity of KRT, assessed up 2 months
  Assess the influence of using NAC in the incidence of the necessity of KRT.
NAC and death | From the post operatory until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 months
  Assess the influence of using NAC in the incidence of death

CONTACTS AND LOCATIONS:
Overall Officials: José J Galvão de Lima, PhD, Principal Investigator — USP InCor
Locations (1):
- José Jayme Galvão de Lima, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We don't have fixed reviewers for our data until our submission for publication

REFERENCES:
- [Background] Spector A. Review: Oxidative stress and disease. J Ocul Pharmacol Ther. 2000 Apr;16(2):193-201. doi: 10.1089/jop.2000.16.193. PMID 10803430
- [Result] Suen WS, Mok CK, Chiu SW, Cheung KL, Lee WT, Cheung D, Das SR, He GW. Risk factors for development of acute renal failure (ARF) requiring dialysis in patients undergoing cardiac surgery. Angiology. 1998 Oct;49(10):789-800. doi: 10.1177/000331979804900902. PMID 9783643
- [Result] Bahar I, Akgul A, Ozatik MA, Vural KM, Demirbag AE, Boran M, Tasdemir O. Acute renal failure following open heart surgery: risk factors and prognosis. Perfusion. 2005 Oct;20(6):317-22. doi: 10.1191/0267659105pf829oa. PMID 16363316